CLINICAL TRIAL: NCT03376594
Title: Efficacy and Safety of Benjakul Extract Capsules and Loratadine for Treatment Allergic Rhinitis Patients (Clinical Trial Phase II)
Brief Title: Benjakul Extract and Loratadine for Treatment Allergic Rhinitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Katanchalee Houngiam, Faculty of Medicine, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-EC-TM-4-183/57
Record Dates: First submitted 2017-06-26; First posted 2017-12-18 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Allergic Rhinitis
Keywords: Benjakul Extract; Allergic Rhinitis; Herbal Medicine
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Loratadine

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator
Masking Description: Grouping uses Randomize controlled trial (RCT) and groups by using Random allocation by means of Simple Randomization as well as using the code with BJK followed by 3 digits (BJK001, BJK002, ...) and treating in double blinding form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benjakul Extract (Active Comparator): Benjakul Extract 100 mg capsule by mouth 3 times a day for 42 days
  Interventions: Drug: Benjakul Extract
- Loratadine (Placebo Comparator): Loratadine 10 mg capsule by mouth 3 times a day for 42 days
  Interventions: Drug: Loratadine

INTERVENTIONS:
Drug: Benjakul Extract — 30 patients taking Benjakul Extract dosage 100 mg capsule 3 times daily. before Breakfast, lunch and dinner for 42 days.
  Other Names: Benjakul remedy
  Arms: Benjakul Extract
Drug: Loratadine — 30 patients taking Loratadine dosage 10 mg capsule 3 times daily. before Breakfast, lunch and dinner for 42 days.
  Other Names: Clarityne
  Arms: Loratadine

SUMMARY:
1. To compare the effectiveness of Benjakul extract capsules at 300 mg per day with Loratadine drug in the treatment of allergic rhinitis patients in small group (Clinical Trial Phase II).
2. To study the safety and side effects of Benjakul extract capsules 300 mg per day and Loratadine drug for allergic rhinitis patients.

DETAILED DESCRIPTION:
1. Group 1consists of 30 patients, taking Benjakul dosage 100 mg or 1 capsule 3 times daily. beforeBreakfast, lunch and dinner.
2. Group 2 consists of 30 patients, taking Loratadine dosage 100 mg 1time daily.Taking drug is as follows

Volunteers will be treated by drugs continuously for a period of six weeks. Taking three times a day 1 tablet before meals (breakfast, lunch, dinner), giving drug based on random.

Volunteers groups receiving Benjakul take 1capsule 3 times daily. Volunteer groups receiving Loratadine take loratadine tablet first 1capsule 1 time daily and then taking placebo once 1 capsule during the day and 1 capsule in the evening.

Patients have to report all the 42 days (6 weeks). The blood and urine samples will be collected and evaluated before the treatment and later following symptoms after 21 and 42 days (3 weeks and 6). Assessment methods to measure the nasal, other of nasal symptoms, assessment of quality of life and overall treatment (Global assessment),Acoustic Rhinometry and tools which are used to evaluate nasal congestion. measuring the narrowest cross-sectional area of the nasal cavity, this tool takes a short time to evaluate and can determine volume of nasal cavity by calculating of the CSA in the nasal cavity. In addition, the researchers areable to check the safety of using medications by taking blood and urine samples to check Hematology CBC, Lipid profile, FBS monitoring of renal function (Renal function test) and liver function tests (Liver Function Tests: LFTs). So, the volunteers must NPO before every blood drawing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 20-70 years
* Patients have history of allergic rhinitis on the basis of Allergic Rhinitis and its Impact on Asthma : ARIA (itching and nasal obstruction, watery nasal discharge, sneezing ,congestion)
* Patients have moderate allergic rhinitis diagnosed by doctor with a minimum TNSS score of 5 points
* No history of disease : heart disease, kidney disease, liver disease, epilepsy,high blood pressure and severe asthma.
* Normal results in blood test, liver and kidney.
* Not pregnant or breastfeeding.
* Body Mass Index (BMI) 18-35 kg / m2 and normal vital signs.
* Volunteers are willing participants.

Exclusion Criteria:

* Volunteers who have taken anti-coagulant and anti-platelet aggregation drugs.
* Patients receiving Intranasal steroids.
* Volunteers who get serious side effect from loratadine : fatigue, headache, dry mouth, drowsiness, nausea, stomach ulcers, rash.
* Volunteers who have side effects from Benjakul drug.
* Volunteers who have a temperature.
* Volunteers participating in other research.
* Volunteers who have severe urticaria and anaphalaxis.
* Volunteers who are immunocompromised or have with severe chronic diseases, such as AIDS.
* Volunteers who have taken Macrolides : erythromycin, clarithromycin, Imidazole (ketoconazole, itraconazole, fluconazole) HIV protease Inhibitors, Other drugs that inhibit the enzyme CYP450: cimetidine,metronidazole,zafirlukast, SSRIS
* Volunteers are using drug which extract QT interval, such as Calcium Channel Blockers (eg bepridil, verapamil), Tricyclic Antidepressant, Cisapride, Quinidine and so on.
* Volunteers have nasal septum perforation or have had sinus surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Nasal clavity | 42 days
  efficacy of the treatments on nasal symptoms and clavity by acoustic rhinometry

SECONDARY OUTCOMES:
Adverse event | 42 days
  Clinical symptoms, Laboratory blood and urine test
Quality of life | 42 days
  quality of life of the patientts by Rhinoconjunctivitis quality of life Questionare (Rcq36)

CONTACTS AND LOCATIONS:
Overall Officials: Katanchalee Houngiam, M.Sc., Principal Investigator — katanchalee01@gmail.com
Locations (1):
- Faculty of Medicine, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
efficacy : (questionnaire, RCQ 36) safety : (Live function test, renal function test, CBC, BP)